CLINICAL TRIAL: NCT01211808
Title: Effect of Diltiazem on the Pharmacokinetics of BMS-914392 and on Heart Rate After Single-dose Administration of BMS-914392 in Healthy Subjects
Brief Title: Effect of Diltiazem on Pharmacokinetics of BMS-914392
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV203-002
Record Dates: First submitted 2010-09-03; First posted 2010-09-30 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (BMS-914832) (Experimental)
  Interventions: Drug: BMS-914832
- Treatment B (BMS-914832 + diltiazem) (Experimental)
  Interventions: Drug: BMS-914832; Drug: Diltiazem

INTERVENTIONS:
Drug: BMS-914832 — Tablets, Oral, 30 mg, once, 1 day
Drug: Diltiazem — Tablets, Oral, 360 mg, once daily, 10 days
  Arms: Treatment B (BMS-914832 + diltiazem)

SUMMARY:
The purpose of this study is to assess the effects of diltiazem on the pharmacokinetics of single-dose BMS-914392 in healthy subjects.

DETAILED DESCRIPTION:
Protocol designed to evaluate the potential for a drug-drug interaction

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy

Exclusion Criteria:

* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Current or history of neurological diseases or psychiatric disorders and cardiovascular diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single dose of BMS-914393 derived from serial measurements of BMS-914392 plasma concentrations | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, and 96 hours after dosing of BMS-914392 alone or in combination with diltiazem

SECONDARY OUTCOMES:
The effect of multiple doses of BMS-914392 on PR, QRS, RR, and QTc intervals derived from serial electrocardiograms (ECGs) | Pre-dose and 0.5 Hr, 1 Hr, 1.5 Hr, 2 Hr, 3 Hr, 4 Hr , 6 Hr, 8 Hr, 12 Hr, 24 Hr after dosing of BMS-914392 alone or in combination with diltiazem
Number of subjects with adverse events as a measure of safety and tolerability of BMS-914392 | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Pra International, Lenexa, Kansas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx